CLINICAL TRIAL: NCT04747951
Title: Total Neoadjuvant Therapy in Rectal Cancer Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Principal Investigator, Rybakov Evgeny, MD, Head of Surgical department of oncoproctology, State Scientific Centre of Coloproctology, Russian Federation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 127872
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; total neoadjuvant therapy; colorectal disease
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy; Radiotherapy; Consolidation Chemotherapy; XELOX; Chemotherapy, Adjuvant

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- total neoadjuvant therapy (Experimental): Total neoadjuvant therapy consisted chemoradiotherapy with capecitabine and nine weeks of consolidation chemotherapy with XELOX prior to surgery and adjuvant therapy if necessary.
  Interventions: Combination Product: Concurrent Chemoradiotherapy; Procedure: TME; Drug: consolidation chemotherapy; Drug: adjuvant chemotherapy
- standard therapy (Active Comparator): Standard therapy (neoadjuvant chemoradiotherapy, surgery, adjuvant chemotherapy)
  Interventions: Combination Product: Concurrent Chemoradiotherapy; Procedure: TME; Drug: adjuvant chemotherapy

INTERVENTIONS:
Combination Product: Concurrent Chemoradiotherapy — 50Gy in 25 fractions to the primary tumor and to mesorectal, presacral,and internal iliac lymph nodes.
  Concurrent chemotherapy:
  Capecitabine 1650 mg/m2/d
  Other Names: Radiotherapy
Procedure: TME — Total mesorectal excision
Drug: consolidation chemotherapy — Intravenous infusion of oxaliplatin (130 mg/m2 over 2 h) on day 1 and oral administration of capecitabine (1000 mg/m2 twice daily) from day 1 to day 14, is repeated every 3 weeks for 3 courses, 3 weeks per course
  Other Names: XELOX; CAPOX
  Arms: total neoadjuvant therapy
Drug: adjuvant chemotherapy — Administration of l-LV (400 mg/m2) and oxaliplatin (85 mg/ m2) by intravenous infusion over 2 h, followed by rapid intravenous infusion (iv) of 5-FU (400 mg/m2) and then slow infusion (civ) of 5-FU (2400 mg/m2 over 46 h), is repeated every 2 weeks for 6-12 cycles
  Other Names: mFOLFOX

SUMMARY:
This is a randomized, controlled, parallel study to determine the efficiency and safety of total neoadjuvant therapy in rectal cancer treatment.

DETAILED DESCRIPTION:
In this randomized, controlled, parallel study we will comparison total neoadjuvant therapy with standard neoadjuvant therapy in rectal cancer treatment. Complete pathological response rate will be the primary endpoint in patients, who will undergoing surgery. In cases of complete clinical response we will provide "watch and wait" approach. Compliance of treatment and oncologic results will be the second endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Have signed an approved informed consent form for the stud;
* Histologically confirmed rectal adenocarcinoma low (cT2-4N0-2M0) or mid rectum (сТ2-T4N1-2M0);

Exclusion Criteria:

* rectal cancer recurrence;
* Primary-multiple tumours of other localizations;
* pelvis radiotherapy in anamnesis;
* pregnancy, breastfeeding;
* distant metastasis;
* ECOG score 3-4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
The rate of complete responses | 3-6 months
  The rate of pathological or clinical complete responses

SECONDARY OUTCOMES:
Rate of R0-resections | immediately after surgery
  Rate of R0-resections
Rate of compliance with radiotherapy and chemotherapy | 6-8 months
  Rate of complications III-VI grade of radiotherapy (RTOG) and chemotherapy (NCI-CTC)
rate of intraoperative and postoperative complications | 0-30 days after surgery
  Frequency and structure of intraoperative and postoperative complications according to the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Rybakov, Dr.Med.Sc, Principal Investigator — Head of Surgical department of oncoproctology
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin ST, Heneghan HM, Winter DC. Systematic review and meta-analysis of outcomes following pathological complete response to neoadjuvant chemoradiotherapy for rectal cancer. Br J Surg. 2012 Jul;99(7):918-28. doi: 10.1002/bjs.8702. Epub 2012 Feb 23. PMID 22362002
- [Background] Zorcolo L, Rosman AS, Restivo A, Pisano M, Nigri GR, Fancellu A, Melis M. Complete pathologic response after combined modality treatment for rectal cancer and long-term survival: a meta-analysis. Ann Surg Oncol. 2012 Sep;19(9):2822-32. doi: 10.1245/s10434-011-2209-y. Epub 2012 Mar 21. PMID 22434243
- [Background] Rodel C, Martus P, Papadoupolos T, Fuzesi L, Klimpfinger M, Fietkau R, Liersch T, Hohenberger W, Raab R, Sauer R, Wittekind C. Prognostic significance of tumor regression after preoperative chemoradiotherapy for rectal cancer. J Clin Oncol. 2005 Dec 1;23(34):8688-96. doi: 10.1200/JCO.2005.02.1329. Epub 2005 Oct 24. PMID 16246976